CLINICAL TRIAL: NCT02263950
Title: A Phase 1/2a Study of LON002 (Sublingual Artemether Spray) in Subjects With Advanced Solid Tumours.
Brief Title: A Phase 1/2a Study of LON002 in Subjects With Advanced Solid Tumours
Acronym: LON002-002
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: LondonPharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LON002-002
Record Dates: First submitted 2014-10-08; First posted 2014-10-15 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Solid Tumours
Keywords: Cancer; Malignant Neoplasm; Artemether; Sublingual; Neoplastic disease; Solid Tumour; Anti-cancer drug; Chemotherapy; LON002
MeSH Terms: conditions — Neoplasms | interventions — Artemether

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LON002 (Experimental): (Artemether sublingual spray)
  Interventions: Drug: Artemether

INTERVENTIONS:
Drug: Artemether — Artemether sublingual spray at 20mg per spray. Dose escalation study design as per protocol; in Phase 1, three dose levels will be given. The Phase 2 dose will be determined from the results of Phase 1. All patients will receive 4 cycles of dosing, 28 days per cycle.
  Other Names: LON002

SUMMARY:
This clinical trial will assess whether a medicine called artemether, currently used at a lower dose to treat malaria, could also be useful in treating cancer. For this trial, the medicine is given in a new way, as a spray under the tongue. This delivery has several advantages, including better absorption into the body and it may be easier for people to take. It will be prescribed to consenting patients with advanced solid tumours, every day for 4 months, either once or twice a day. (For this study 'advanced tumour' will mean there are no other effective standard therapy options available to the patient).

The dose will be decided in Phase 1 of the study by initially testing 3 different doses of the medicine in up to 21 different cancer patients, to make sure it is not too toxic or causes any side effects.

After this, the highest safe dose identified in the first phase will be tested in up to 66 cancer patients in Phase 2 of the study, to see if the medicine is able to reduce the size of their tumour or slow down its growth.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of 18 years or older at the Screening Visit.
2. Histologic and/or cytologically confirmed diagnosis of solid tumour with clinical and imaging evidence that the tumour is advanced and for whom there is no effective standard therapy available.
3. At least one evaluable tumour that is at least 10 mm by computerised tomography (CT) scan or magnetic resonance imaging (MRI) at the pre-treatment stage
4. At least one prior systemic anti-cancer treatment and disease that is refractory or progressive following treatment.
5. Eastern Co operative Oncology Group (ECOG) performance ≤ 2.
6. An adequate renal, liver and bone marrow function.
7. Women of child bearing potential (WOCBP) must have a negative pregnancy test before the start of treatment.
8. Sexually active women of childbearing potential must be using an acceptable form of contraception, as detailed in the protocol.
9. Male subjects must have had a successful vasectomy (confirmed azoospermia) or they and their female partner must meet the criteria defined in the protocol (i.e., not of childbearing potential or practicing highly effective contraception throughout the study period and for 30 days after study drug discontinuation). Those with partners using hormonal contraceptives must also be using an additional approved method of barrier contraception.
10. Expected life expectancy > 4 months.

Exclusion Criteria:

1. Unwillingness or inability to provide informed consent.
2. Any evidence of severe or uncontrolled systemic diseases, infection or laboratory finding that in the view of the Investigator makes it undesirable for the patient to participate in the trial.
3. Allergic to artemether or other artemisinin derivatives or any of the components of the sublingual formulation.
4. Pregnancy or lactation.
5. Subject had major surgery or significant traumatic injury within 4 weeks of start of study drug; subject has not recovered from the side effects of any major surgery (defined as requiring general anaesthesia) or subject might require major surgery during the course of the study.
6. Subject has had anti-cancer treatment within 4 weeks of start of study drug, excluding small field palliative irradiation which may be performed up to 2 weeks prior to start of study drug.
7. Subject has had prior treatment with any investigational drug within the preceding 4 weeks before study start.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Determination of the Recommended Phase 2 Dose (RP2D) to be used in Phase 2a of the study | 28 days
Number (%) of patients with clinical benefit in Phase 2a | 16 weeks
  * Complete or partial response at any time based on imaging
  * Stable disease at 16 weeks (4 cycles); and/or
  * Reduction of validated biomarkers

SECONDARY OUTCOMES:
Number of subjects with Dose limiting toxicities | 16 weeks
Time to progression (TTP), progression free survival (PFS) and overall survival (OS). | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Debashis Sarker, MD, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust; Mazhar Ajaz, MD, Principal Investigator — Royal Surrey County Hospital NHS Trust; Daryl Bendel, MD, Study Director — Xidea Solutions Ltd.
Locations (2):
- United Kingdom (2):
  - The Royal Surrey County Hospital, Guildford, Surrey
  - Guy's and St Thomas NHS Foundation Trust, London